CLINICAL TRIAL: NCT02850185
Title: Adjuvant Therapy for Severe COPD Patients in the Stable Phase by an Oxyhydrogen Generator With Nebulizer: A Multi-centric, Randomized, Parallel-control and Double-blinded Clinic Study
Brief Title: Adjuvant Therapy for Severe COPD Patients in the Stable Phase by an Oxyhydrogen Generator With Nebulizer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Asclepius Meditec Inc. (Industry)
Collaborators: West China Hospital (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); The Second Hospital of Hebei Medical University (Other); Tianjin Medical University General Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Ze-guang Zheng, Clinical Professor, Shanghai Asclepius Meditec Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ZZheng
Record Dates: First submitted 2016-07-22; First posted 2016-07-29 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-04

CONDITIONS: COPD
Keywords: COPD; hydrogen
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Nebulizers and Vaporizers; Oxygen Inhalation Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oxyhydrogen (Experimental): conventional treatment (bronchodilator (LABA,LAMA) with or without ICS)+ hydrogen/ oxygen inhaled
  Interventions: Device: oxyhydrogen; Drug: Conventional treatment
- oxygen (Experimental): conventional treatment (bronchodilator (LABA,LAMA) with or without ICS)+ oxygen inhaled
  Interventions: Device: Oxygen; Drug: Conventional treatment

INTERVENTIONS:
Device: oxyhydrogen — Hydrogen/oxygen mixed gas inhaled(proportion 2:1),3 L/min . 1 hour each time,twice a day(BID).Test Duration is three months.
  Other Names: Oxyhydrogen generator with nebulizer
  Arms: oxyhydrogen
Device: Oxygen — oxygen inhaled,3 L/min . 1 hour each time,twice a day(BID).Test Duration is three months.
  Other Names: Medical molecular sieve oxygenerator
  Arms: oxygen
Drug: Conventional treatment — Bronchodilator (LABA,LAMA) with or without ICS.Conventional treatment is invariable with which was given to COPD patients in 3 months before the study.
  Other Names: medication treatment

SUMMARY:
The purpose for this study is to determine safety and effectiveness of the oxyhydrogen generator with nebulizer through an adjuvant therapy for the severe COPD patients in the stable phase.

DETAILED DESCRIPTION:
In this study, severe COPD patients in stable phase who were included in both treatment and control groups, administered randomly oxyhydrogen generator with nebulizer (treatment group) or oxygen Nebulizer Machine （control group ）for adjuvant therapy. The therapeutic outcomes in both treatment and control groups are analyzed and evaluated to verify safety and effectiveness of the test product.This study is a multi-center, randomized, double-blind study. The trial lasted for 3 months. The curative effect was observed for subjects in the second week, first month, second month and third month respectively as the observing time point. Total patients which are planned to be included are 140 cases, where, 70 cases in the treatment group and control group respectively are distributed in 5 clinical hospitals.

ELIGIBILITY:
Inclusion Criteria:

1. It conforms to the diagnostic criteria of chronic obstructive pulmonary diseases (COPD): (PFT)The percentage of forced expiratory volume in forced vital capacity in one second after inhaling vasodilator (FEV1 / FVC% < 70%);
2. Classification of COPD severity by pulmonary function: The criterion for this study is Severe: FEV1/FVC<0.70, and FEV1< 50% expected value after pulmonary function was examined by taking bronchodilator.
3. More than 40 years old and have normal ability to judge independently; men and women are not limited;
4. Living in the vicinity of the test centre in the past six months; -

Exclusion Criteria:

* 1) Those who have acute exacerbation in the past 4 weeks; 2) Lung disease history: Excluding the history of other lung diseases except combined COPD, such as combined pulmonary tuberculosis and diffuse pan-capillary bronchiolitis, pneumonia, pneumothorax, pleural effusion, pulmonary embolism, etc.

  3) Those who suffer infectious diseases such as hepatitis A, hepatitis B, AIDS and tuberculosis or connective tissue diseases in the active period; 4) Those who suffer high fever, as well as various local or systemic infections (including respiratory, urinary and reproductive system, digestive system, sepsis, etc.), severe infection, especially lung infection found by CT examination; 5) Those who have limited ability to understand and poor compliance; do not have the legal capacity or limited legal capacity; participated in other clinical trials in the first 3 months when they were included in the groups; mental or physical disability; 6) Those who were difficult to make an exact evaluation on safety and effectiveness of products; 7) The women in pregnancy and lactation, as well as the women at childbearing age who don't agree to take effective contraceptive measures during the study period; 8) Those who have abnormal heart function and thrombophlebitis; 9) Those who are known and can't stand the oxygen and hydrogen inhalation; 10) Those who are suffered from primary diseases in important visceral organs and systems, such as stroke, severe hypertension, gastric ulcer, uncontrolled diabetes, malignant tumor, liver and kidney failure, and severe heart disease history (acute myocardial infarction, congestive heart failure and other heart diseases in the acute phase); 11) Cancer in progressive stage as well as undetermined masses found in the treatment; 12) Those who have one or more lobectomy history; 13) Those who are suspected to have or really have alcohol and drug abuse history; 14) Those whose AST and ALT≥120U/L, Ccr≤50ml/min; who have shock or unstable hemodynamics; 15) Those who are considered not to participate in clinical trials by the investigators.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2016-07-15; Primary Completion 2020-07-21 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in dyspnea index score (mMRC score) at 3 months | baseline and 3 months

SECONDARY OUTCOMES:
Change from Baseline in St George's respiratory questionnaire (SGRQ score) at 3 months | baseline and 3 months
Change from Baseline in Six minute walk distance at 3 months | baseline and 3 months
Change from Baseline in Pulmonary artery pressure measured by heart color Doppler ultrasound at 3 months | baseline and 3 months
Change from Baseline in Forcibly vital capacity(FVC) at 3 months | baseline and 3 months
Change from Baseline in First second forcibly expiration quantity(FEV1) at 3 months | baseline and 3 months
Change from Baseline in mean maximum expiratory flow(MMEF) at 3 months | baseline and 3 months
Change from Baseline in Residual volume(RV) at 3 months | baseline and 3 months
Change from Baseline in Serum interleukin-6(IL-6) at 3 months | baseline and 3 months
Change from Baseline in Serum interleukin-8( IL - 8) at 3 months | baseline and 3 months
Change from Baseline in Serum tumor necrosis factor-a(TNF-a) at 3 months | baseline and 3 months
Change from Baseline in Serum malondialdehyde (MDA) at 3 months | baseline and 3 months
Change from Baseline in Serum 8-isoprostane at 3 months | baseline and 3 months
Change from Baseline in Arterial oxygen tension (PaO2) at 3 months | baseline and 3 months
Change from Baseline in carbon dioxide arterial tension (PaCO2) at 3 months | baseline and 3 months
number of participants with adverse events | up to 3 months
  the adverse events including chest distress,wheezing,cough,heartbeat accelerating,abdominal pain,diarrhea,nausea,vomiting,cardiac,liver, renal toxicity , etc.

CONTACTS AND LOCATIONS:
Overall Officials: Zhong N Shan, academician, Study Chair — First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
the main evaluation index and the secondary evaluation index of all participants will be share in 3 months after the end of this study.

REFERENCES:
- [Background] Ohsawa I, Ishikawa M, Takahashi K, Watanabe M, Nishimaki K, Yamagata K, Katsura K, Katayama Y, Asoh S, Ohta S. Hydrogen acts as a therapeutic antioxidant by selectively reducing cytotoxic oxygen radicals. Nat Med. 2007 Jun;13(6):688-94. doi: 10.1038/nm1577. Epub 2007 May 7. PMID 17486089
- [Background] Liu FT, Xu SM, Xiang ZH, Li XN, Li J, Yuan HB, Sun XJ. Molecular hydrogen suppresses reactive astrogliosis related to oxidative injury during spinal cord injury in rats. CNS Neurosci Ther. 2014 Aug;20(8):778-86. doi: 10.1111/cns.12258. Epub 2014 Mar 31. PMID 24685114
- [Background] Kohama K, Yamashita H, Aoyama-Ishikawa M, Takahashi T, Billiar TR, Nishimura T, Kotani J, Nakao A. Hydrogen inhalation protects against acute lung injury induced by hemorrhagic shock and resuscitation. Surgery. 2015 Aug;158(2):399-407. doi: 10.1016/j.surg.2015.03.038. Epub 2015 May 14. PMID 25983276
- [Background] Nakao A, Toyoda Y, Sharma P, Evans M, Guthrie N. Effectiveness of hydrogen rich water on antioxidant status of subjects with potential metabolic syndrome-an open label pilot study. J Clin Biochem Nutr. 2010 Mar;46(2):140-9. doi: 10.3164/jcbn.09-100. Epub 2010 Feb 24. PMID 20216947
- [Background] Xiao M, Zhu T, Wang T, Wen FQ. Hydrogen-rich saline reduces airway remodeling via inactivation of NF-kappaB in a murine model of asthma. Eur Rev Med Pharmacol Sci. 2013 Apr;17(8):1033-43. PMID 23661516
- [Background] Ning Y, Shang Y, Huang H, Zhang J, Dong Y, Xu W, Li Q. Attenuation of cigarette smoke-induced airway mucus production by hydrogen-rich saline in rats. PLoS One. 2013 Dec 20;8(12):e83429. doi: 10.1371/journal.pone.0083429. eCollection 2013. PMID 24376700
- [Background] Zheng J, Liu K, Kang Z, Cai J, Liu W, Xu W, Li R, Tao H, Zhang JH, Sun X. Saturated hydrogen saline protects the lung against oxygen toxicity. Undersea Hyperb Med. 2010 May-Jun;37(3):185-92. PMID 20568549
- [Background] Kawamura T, Wakabayashi N, Shigemura N, Huang CS, Masutani K, Tanaka Y, Noda K, Peng X, Takahashi T, Billiar TR, Okumura M, Toyoda Y, Kensler TW, Nakao A. Hydrogen gas reduces hyperoxic lung injury via the Nrf2 pathway in vivo. Am J Physiol Lung Cell Mol Physiol. 2013 May 15;304(10):L646-56. doi: 10.1152/ajplung.00164.2012. Epub 2013 Mar 8. PMID 23475767
- [Background] Huang CS, Kawamura T, Peng X, Tochigi N, Shigemura N, Billiar TR, Nakao A, Toyoda Y. Hydrogen inhalation reduced epithelial apoptosis in ventilator-induced lung injury via a mechanism involving nuclear factor-kappa B activation. Biochem Biophys Res Commun. 2011 May 6;408(2):253-8. doi: 10.1016/j.bbrc.2011.04.008. Epub 2011 Apr 5. PMID 21473852
- [Background] Sun Q, Cai J, Liu S, Liu Y, Xu W, Tao H, Sun X. Hydrogen-rich saline provides protection against hyperoxic lung injury. J Surg Res. 2011 Jan;165(1):e43-9. doi: 10.1016/j.jss.2010.09.024. Epub 2010 Oct 15. PMID 21067781